CLINICAL TRIAL: NCT00457340
Title: Cholesterol Lowering and Arrhythmia Recurrences After Internal Defibrillator Implantation (CLARIDI)
Brief Title: Atorvastatin For The Reduction Of Ventricular Arrhythmias
Acronym: CLARIDI
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A2581020
Record Dates: First submitted 2007-04-04; First posted 2007-04-06 (Estimated); Last update posted 2021-02-18 (Actual); Status verified 2021-02

CONDITIONS: Arrhythmia
Keywords: Tachycardia, Ventricular; Ventricular Fibrillation
MeSH Terms: conditions — Arrhythmias, Cardiac; Tachycardia, Ventricular; Ventricular Fibrillation | interventions — Atorvastatin

INTERVENTIONS:
Drug: Atorvastatin 80mg

SUMMARY:
To assess in patients with CAD [coronary artery disease] and an implantable defibrillator the effect of atorvastatin 80 mg versus placebo on the first recurrence of a ventricular arrhythmia (ventricular tachycardia or ventricular fibrillation requiring ICD [implantable cardioverter defibrillator] intervention) within one year after randomization.

ELIGIBILITY:
Inclusion Criteria:

* Eligible subjects were male or female subjects, age >18 years, with clinically documented coronary artery disease and life-threatening ventricular arrhythmias who met the following criteria:
* Were scheduled for an ICD implantation or had an ICD implantation within 1 month, according to the class I American College of Cardiology/American Heart Association (ACC/AHA) practice guidelines for ICD therapy

OR

* Were already treated with an ICD for a class I ACC/AHA indication for more than one month, provided they received at least one appropriate ICD intervention (shock or antitachycardia pacing (ATP) for ventricular tachycardia or ventricular fibrillation) during the preceding six months

Exclusion Criteria:

* Patients with ventricular arrhythmias in the acute phase of myocardial infarction (first 48 hours).
* Patients with incessant ventricular tachycardia.
* Patients with ventricular arrhythmias without underlying coronary artery disease.
* Patients with a transient or reversible cause of ventricular arrhythmias (including significant electrolyte disturbances or drug induced proarrhythmia).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220
Dates: Start 2000-02; Study Completion 2004-09 (Actual)

PRIMARY OUTCOMES:
To assess in patients with CAD and an implantable defibrillator the effect of atorvastatin 80 mg versus placebo on the first recurrence of a ventricular arrhythmia after randomisation.

SECONDARY OUTCOMES:
Combined total mortality and major cardiovascular events.
Major cardiovascular events include acute myocardial infarction, stroke and PTCA [percutaneous coronary angioplasty] (with or without stenting) or CABG [coronary artery bypass graft] (CABG already foreseen at the moment of randomization).
Total number of appropriate ICD interventions for ventricular arrhythmias and total number of episodes of electrical storm.
An episode of electrical storm is defined as the occurrence within 24 hours of three or more ventricular arrhythmias requiring ICD intervention.
Combined total mortality, major cardiovascular events and total number of appropriate ICD interventions for ventricular arrhythmias.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (10):
- Belgium (7):
  - Pfizer Investigational Site, Aalst
  - Pfizer Investigational Site, Antwerp
  - Pfizer Investigational Site, Bruges
  - Pfizer Investigational Site, Edegem
  - Pfizer Investigational Site, Ghent
  - Pfizer Investigational Site, Hasselt
  - Pfizer Investigational Site, Leuven
- Greece (3):
  - Pfizer Investigational Site, Athens
  - Pfizer Investigational Site, Crete
  - Pfizer Investigational Site, RIO Patra

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A2581020&StudyName=Atorvastatin+For+The+Reduction+Of+Ventricular+Arrhythmias